CLINICAL TRIAL: NCT02361346
Title: Safety, Pharmacodynamics and Efficacy of MT-3724 for the Treatment of Patients With Relapsed or Refractory DLBCL
Brief Title: Safety, PD & Efficacy of MT-3724 for the Treatment of Patients With Relapsed or Refractory DLBCL
Acronym: MT-3724NHL001
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision following clinical hold
Sponsor: Molecular Templates, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-3724_NHL_001
Record Dates: First submitted 2015-02-03; First posted 2015-02-11 (Estimated); Results first posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-07

CONDITIONS: Non-Hodgkin's B-cell Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Small Lymphocytic Leukemia; Diffuse Large B Cell Lymphoma; Blood Cancer; Hematological Malignancy
Keywords: CD20; immunotoxin; NHL; non-Hodgkin's lymphoma; lymphoma; cancer; antibodies; immunotherapy; safety; pharmacokinetics; maximum tolerated dose; MT-3724; relapsed; refractory; leukemia; CLL; SLL; DLBCL; efficacy
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Hematologic Neoplasms; Lymphoma, Non-Hodgkin; Lymphoma; Neoplasms; Recurrence; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Part 1: Cohort 1 - 5 Micrograms/Kilogram/Dose (mcg/kg/Dose) (Experimental): Part 1: MT-3724 5 mcg/kg/dose IV for 6 doses over 12 days, followed by dose escalations (Part 1) until recommended phase 2 dose of MT-3724 is determined
  Interventions: Drug: MT-3724 Phase 1
- Part 1: Cohort 2- 10 mcg/kg/Dose (Experimental): Part 1: MT-3724 10 mcg/kg/dose IV for 6 doses over 12 days, followed by dose escalations (Part) until recommended phase 2 dose of MT-3724 is determined
  Interventions: Drug: MT-3724 Phase 1
- Part 1: Cohort 3- 20 mcg/kg/Dose (Experimental): Part 1: MT-3724 20 mcg/kg/dose IV for 6 doses over 12 days, followed by dose escalations (Part 1) until recommended phase 2 dose of MT-3724 is determined
  Interventions: Drug: MT-3724 Phase 1
- Part 1: Cohort 4- 50 mcg/kg/Dose (Experimental): Part 1: MT-3724 50 mcg/kg/dose IV for 6 doses over 12 days, followed by dose escalations (Part 1) until recommended phase 2 dose of MT-3724 is determined
  Interventions: Drug: MT-3724 Phase 1
- Part 1: Cohort 5- 100 mcg/kg/Dose (Experimental): Part 1: MT-3724 100 mcg/kg/dose IV for 6 doses over 12 days, followed by dose escalations (Phase 1) until recommended phase 2 dose of MT-3724 is determined
  Interventions: Drug: MT-3724 Phase 1
- Part 1: Cohort 6- 75 mcg/kg/Dose (Experimental): Part 1b: MT-3724 75 mcg/kg/dose IV for 6 doses over 12 days of 21-Day cycle for up to 4 additional cycles to explore safety, tolerability and tumor response to repeat doses of MT-3724 (subject will continue with dose that was tolerated in the Part 1 portion of the study)
  Interventions: Drug: MT-3724 Phase 1
- Part 2: Cohort 7- MTD Expansion Cohort (Experimental): Part 2: MT-3724 IV for 6 doses administered within 14 days of 21-Day cycle up to 6 Cycles. If the Subject exhibits stable disease or PR after end of Cycle 6 and investigator determines ratio is favorable, treatment with MT- 3724 may be continued for up to additional 6 cycles.
  Interventions: Drug: MT-3724 Phase 1; Drug: MT-3724 Phase 2
- Part 3: All MT-3724 Treated Participants (Experimental): Part 3: MT-3724 IV 50 µg/kg/dose administered on Days 1, 3, 5, 8, 10, and 12 of each 21-day cycle. Treatment will continue until death, disease progression, unacceptable toxicity, withdrawal of consent, or another reason for withdrawal, or until study discontinuation
  Interventions: Drug: MT-3724 Phase 2
- Part 4: All MT-3724 Treated Participants (Experimental): Part 4: In this arm, subjects were planned to receive all doses of MT-3724 as IV infusion as confirmed in Part 3.
  Interventions: Drug: MT-3724 Phase 2

INTERVENTIONS:
Drug: MT-3724 Phase 1 — Intravenous dosing Days 1, 3, 5, 8, 10 and 12; MT-3724 infusion over 2 hours on each dosing day over 28 day initial cycle and then 21 week repeat cycles for up to 5 total cycles.
  Arms: Part 1: Cohort 1 - 5 Micrograms/Kilogram/Dose (mcg/kg/Dose); Part 1: Cohort 2- 10 mcg/kg/Dose; Part 1: Cohort 3- 20 mcg/kg/Dose; Part 1: Cohort 4- 50 mcg/kg/Dose; Part 1: Cohort 5- 100 mcg/kg/Dose; Part 1: Cohort 6- 75 mcg/kg/Dose; Part 2: Cohort 7- MTD Expansion Cohort
Drug: MT-3724 Phase 2 — Intravenous dosing on Days 1, 3, 5, 8, 10 and 12; MT-3724 infusion over 1 hour on each dosing day over 21 day cycle up to 6 cycles and then can be continued for 6 additional cycles.
  Arms: Part 2: Cohort 7- MTD Expansion Cohort; Part 3: All MT-3724 Treated Participants; Part 4: All MT-3724 Treated Participants

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of MT-3724 in subjects with relapsed or refractory B-Cell NHL or relapsed and refractory CLL (Part 1 only) and relapsed and refractory DLBCL (Part 2 and Part 3). Part 3 evaluates the efficacy of MT-3724.

DETAILED DESCRIPTION:
This is a three-part Phase 2 study

Part 1: (MT-3724 Dose Escalation) Define the maximum tolerated dose (MTD) of MT-3724 [Completed]

Part 2: (MTD Expansion Cohort) Confirm the safety and tolerability of the MTD of MT-3724 in the MTD Expansion Cohort.

Part 3: (Phase 2 MTD Expansion Cohort) Determine the efficacy of MT-3724 as monotherapy in subjects with relapsed or refractory DLBCL based on the overall response rate (ORR) by the revised Lugano Classification for Lymphoma adjusted according to LYRIC.

It is anticipated that up to 100 patients will be enrolled in Part 3. Treatment will continue for up to six 21 days cycles. If the subject exhibits SD, CR or PR after the end of Cycle 6 and the investigator determines that the benefit-risk ratio is favorable, then the treatment with MT-3724 may be continued after discussion with the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be informed about the study and fully consent to participation as demonstrated by signing the written ICF before any screening procedure.
* Male and female participants >= 18 years of age at the time of informed consent.
* Participants must have relapsed or refractory Diffuse large B cell lymphoma (DLBCL) according to the Revised European American Lymphoma/World Health Organization classification. Participants must have proof of cluster of differentiation 20 plus (CD20+) DLBCL, based on either:

  * a. historical biopsies (obtained with diagnosis of relapsed or refractory disease), or
  * b. fresh biopsies
  * c. bone marrow biopsy, excisional lymph node biopsy, and core biopsy of any involved organ are all acceptable methods; Fine Needle Aspirate is not acceptable.
* Participants must have received at least 2 standard of care (SoC) regimens (including anti-CD20 antibody therapy) appropriate for DLBCL treatment.

  * a. Participants whose prior therapy includes chimeric antigen receptor T-cell (CAR-T-cell) therapy are eligible.
  * b. Participants who underwent stem cell transplant (SCT) > 100 days for autologous SCT or > 180 days for allogeneic SCT before study drug administration.
  * c. Participants who have been ineligible for SoC DLBCL treatments may be eligible at the investigator's discretion, upon sponsor approval.
* Participants must have at least 1 bi-dimensional tumor lesion at screening that is measurable by computerized tomography (CT) and/or magnetic resonance imaging (MRI) according to the Lugano criteria. Bi-dimensionally measurable tumor lesion by CT and/or MRI is defined as longest diameter of > 1.5 centimeters (cm) for lymph nodes and > 1.0 cm for extranodal disease.
* Participants must have life expectancy of > 3 months from the start of treatment.
* Participants must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Participants must have met ALL the following laboratory criteria:

  * a. absolute neutrophil count (ANC) >= 1.0 × 10^9 cells per liter with no myeloid growth factors (granulocyte colony-stimulating factor [G-CSF] or granulocyte-macrophage colony-stimulating factor preparations) administered within 2 weeks of Cycle 1 Day 1.
  * b. platelet count >= 50 × 10^9 cells per liter with no Thrombopoietin-receptor agonists agents or platelet transfusions given within 2 weeks of Cycle 1 Day 1.
  * c. hemoglobin >= 8.0 grams per deciliter (g/dL) with no erythropoietin stimulating agents or peripheral red blood cell (PRBC) transfusions within 2 weeks of Cycle 1 Day 1
  * d. creatinine clearance (CLcr) to be >= 50 milliliter per minute (ml/min) either measured or estimated using the Cockcroft-Gault formula.
  * e. total bilirubin (or direct bilirubin for patients with Gilbert's disease < 1.5 × upper limit of normal (ULN)
  * f. alanine transaminase (ALT) ≤ 3.0 × ULN (or <= 5.0 x ULN if liver involvement).
  * g. aspartate aminotransferase (AST) <= 3.0 × ULN (or <= 5.0 x ULN if liver involvement).
  * h. international normalized ratio (INR) or prothrombin time (PT) <= 1.5 x ULN (unless on therapeutic anticoagulants).
  * i. Activated partial thromboplastin time <= 1.5 x ULN (unless on therapeutic anticoagulants).
* Have adequate serum albumin, as determined by: a. albumin >= 3.0 g/dL.
* QT interval correction for heart rate using Fridericia's formula (QTcF) <= 480 milliseconds determined as the average of 3 QTcF values from the triplicate electrocardiogram (ECG) obtained at screening.
* Women of reproductive potential must have a negative highly sensitive pregnancy test within 72 hours before the start of treatment. Women who are postmenopausal or permanently sterilized (eg, tubal occlusion, hysterectomy, bilateral salpingectomy) may be considered as not of reproductive potential.
* Participants of reproductive potential must agree either to abstain continuously from heterosexual intercourse or to use a highly effective birth control method from signing the informed consent until the short term follow-up (STFU) visit for females and until 90 days after the last dose of MT-3724 for males.
* Participants must be able to comply with all study-related procedures and medication use.

Exclusion Criteria

Prior or Current Therapies

* Received any amount of anti-CD20 monoclonal antibodies (mAbs) within the following periods before the start of treatment:

  * a. Rituximab (Rituxan®/MabThera® or rituximab biosimilar): within 84 days (12 weeks); if a participant has received rituximab within 37 weeks before the start of treatment, then serum rituximab level must be negative (< 500 nanograms per milliliter [ng/mL]) at screening.
  * b. Obinutuzumab (Gazyva®/Gazyvaro®): 184 days c. Ofatumumab (Arzerra®): 88 days d. Any other anti-CD20 agents (eg, investigational agents), the washout period is 5 half-lives. The investigator must contact the medical monitor to discuss the most Compound: MT-3724 appropriate washout for non-approved CD20-targeting agents, where the half-life (t1/2) is not known.
* Received approved or investigational treatment for DLBCL within 4 weeks before the start of treatment. For small molecules (MW < 0.9 kilodaltons [kDa]), the washout is 5 half-lives or at least 2 weeks. Radioimmunoconjugates are excluded within 12 weeks before the start of treatment.
* Received radiation therapy to tumor lesions that would serve as target lesions (measurable disease) within 4 weeks before the start of treatment, unless the lesion exhibited objective progression between radiation therapy and screening according to the Lugano Classification

  o a. Palliative radiation therapy to non-target lesions may be permitted at the investigator's discretion after consultation with the medical monitor and sponsor.
* Require the use of systemic immune modulators during study treatment:

  * a. Systemic immune modulators include, but are not limited to, systemic corticosteroids at doses > 20 milligrams per day (mg/day) of prednisone equivalent, cyclosporine and tacrolimus.
  * b. The use of non-steroidal anti-inflammatory drugs (NSAIDS) is permitted.
* Received any live vaccines within 4 weeks before the start of treatment.
* Prior treatment with MT-3724.

Medical History

* Current evidence of Common Terminology Criteria for Adverse Events (CTCAE) Grade > 1 toxicity (due to prior anticancer therapy) before the start of treatment, except for hair loss and those Grade 2 toxicities listed as permitted in other eligibility criteria.
* Current evidence of significant (CTCAE Grade ≥ 2) infection or wound within 4 weeks before the start of treatment. a. Participants with Grade 2 infection that has stabilized or improved with oral anti-infectives before the start of treatment may be eligible at the sponsor's discretion.
* Known or suspected hypersensitivity to the study drug or excipients contained in the study drug formulation.
* Current evidence of hypersensitivity or other underlying illness requiring systemic corticosteroids at doses > 20 mg/day prednisone equivalent.
* Current evidence of uncontrolled human immunodeficiency syndrome (HIV), hepatitis B virus (HBV) or /hepatitis C virus (HCV) at screening. Serology testing is not required if seronegativity is documented in the medical history, and if there are no clinical signs suggestive of HIV or hepatitis infections, or suspected exposure. The following exceptions apply for participants with positive viral serology:

  * a. Participants with HIV and an undetectable viral load and CD4+ T-cell (CD4+) counts >= 350 cells per milliliter may be enrolled, but must be taking appropriate opportunistic infection prophylaxis, if clinically relevant.
  * b. Participants with positive HBV serology are eligible if they have an undetectable viral load and the participant will receive antiviral prophylaxis for potential HBV reactivation per institutional guidelines.
  * c. Participants with positive HCV serology are eligible if quantitative polymerase chain reaction (PCR) for plasma HCV ribonucleic acid (RNA) is below the lower limit of detection. Concurrent antiviral HCV treatment per institutional guidelines is allowed.
* Current evidence of incomplete recovery from surgery or radiotherapy before start of treatment, or planned surgery or radiotherapy from the start of treatment until the end of treatment (EoT) visit, except minor elective surgery deemed acceptable by the investigator or palliative radiation therapy to non-target lesions.
* History of cardiovascular, renal, hepatic or any other disease within 3 months before the start of treatment that in the investigator's opinion, may increase the risks associated with study participation or require treatments that may interfere with the conduct of the study or the interpretation of study results.
* History or current evidence of neoplastic disease that is histologically distinct from NHL, except cervical carcinoma in situ, superficial noninvasive bladder tumors, curatively treated Stage I-II non-melanoma skin cancer. Participants with prior, curatively treated cancer > 2 years ago before the start of treatment can be enrolled.
* Current evidence of new or growing brain or spinal metastases during screening. Participants with known brain or spinal metastases may be eligible if they:

  * a. Had radiotherapy or another appropriate therapy for the brain or spinal metastases; concurrent prophylactic treatment is allowed
  * b. Neurologic symptoms must be stable and no worse than Grade 2
  * c. Have evidence of stable brain or spinal disease on CT or MRI scan obtained within 4 weeks before signing the informed consent and compared with prior imaging results
  * d. Do not require steroid therapy (or, if applicable, have been stable on dose of no more than prednisone 20 mg/day or equivalent by C1D1)
* Women who are pregnant or breastfeeding.
* History of non-adherence to the schedule of procedures or medication use. 18. Current evidence of Graft vs Host Disease
* History or current evidence of significant cardiovascular disease including, but not limited to, the following conditions:

  * a. Unstable angina (symptoms of angina at rest) or new-onset angina within 3 months before the start of treatment.
  * b. Arterial thrombosis or pulmonary embolism within 3 months before the start of treatment.
  * c. Myocardial infarction or stroke within 3 months before the start of treatment.
  * d. Pericarditis (any CTCAE grade), pericardial effusion (CTCAE Grade >= 2), non-malignant pleural effusion (CTCAE Grade ≥ 2) or malignant pleural effusion (CTCAE Grade >= 3) within 3 months before the start of treatment with MT-3724.
  * e. Congestive heart failure (New York Heart Association [NYHA] Class III or IV) at screening or left ventricular ejection fraction (LVEF) <= 45 percent (%), assessed by echocardiogram (ECHO) or multigated acquisition (MUGA) scan within 1 month before starting study treatment (inclusion of participants with LVEF between 40% to 45% should be discussed with the medical monitor and approved by the sponsor). (ECHO or MUGA performed within 6 months before screening and at least 28 days after the last cancer therapy is acceptable provided the participant has not received any potentially cardiotoxic agents since then).
  * f. Cardiac arrhythmia requiring anti-arrhythmic therapy at screening. Participants receiving digoxin, calcium channel blockers, or beta-adrenergic blockers are eligible at the investigator's discretion after consultation with medical monitor and sponsor if the dose has been stable for >= 2 weeks before the start of treatment with MT-3724. Participants with sinus arrhythmia and infrequent premature ventricular contractions are eligible at the investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (16):
  - University of Arizona, Tucson, Arizona
  - Innovative Clinical Research Institute, LLC, Whittier, California
  - 21st Century Oncology - Jacksonville, Jacksonville, Florida
  - Orlando Health, Inc., Orlando, Florida
  - BRCR Medical Center, Plantation, Florida
  - ASCLEPES Research Centers, Weeki Wachee, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - University of Illinois, Cancer Center, Chicago, Illinois
  - Healthcare Research Network III, LLC, Tinley Park, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Norton Healthcare, Inc, Louisville, Kentucky
  - New York University Langone Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - UT Health San Antonio Cancer, San Antonio, Texas
- Belarus (2):
  - Grodno University Hospital, Grodno
  - Minsk City Clinical Oncology Center, Minsk
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Montreal Oncology Research, Québec
- LLC ARENSIA Exploratory Medicine, Tbilisi, Georgia
- Israel (3):
  - Rabin Medical Center, Davidoff Cancer Center, Hemato-Oncology Institute, Petah Tikva
  - Chaim Sheba Medical Center, Department of Hematology, Ramat Gan
  - The Tel Aviv Sourasky Medical Center, Department of Hematology and Bone Marrow Transplantation, Tel Aviv
- ARENSIA Exploratory Medicine,, Chisinau, Moldova
- Poland (6):
  - Maria Sklodowska-Curie National Institute of Oncology - National Research Institute, Gliwice
  - University Hospital in Krakow, Teaching Unit of the Hematology Department, Krakow
  - Frederic Chopin Provincial Teaching Hospital, Teaching Department of Hematology, Rzeszów
  - Our Doctor Clinical Trials Center, Torun
  - Institute of Hematology and Transfusion Medicine, Department of Hematology, Warsaw
  - Jan Mikulicz Radecki University Hospital in Wroclaw, Department and Clinic of Hematology, Blood Neoplasms and Bone Marrow Transplantation, Wroclaw
- Serbia (2):
  - Clinical Center Kragujevac, Clinic of Hematology, Kragujevac
  - Clinical Center of Vojvodina, Clinic of Hematology, Novi Sad
- Spain (4):
  - Catalan Institute of Oncology (ICO) - Hospital Duran i Reynals, Department of Clinical Hematology, Barcelona
  - University Hospital Vall d'Hebron (HUVH), Department of Hematology, Barcelona
  - Hospital Universitario QuironSalud Madrid, Madrid
  - University Hospital Virgen del Rocio (HUVR), Department of Hematology, Seville
- Medical Center of Limited Liability Company "Medical Centre Named by Academician Yurii Spizhenko, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This 4-part study evaluated safety, pharmacodynamics and efficacy of MT-3724 in participants with relapsed or refractory diffuse large B-cell lymphoma (DLBCL). Part 1 was multiple ascending dose study and Parts 2, 3 and 4 were multi-center, multinational, open-label, single-arm evaluation of MT-3724 administered as monotherapy in repeat doses.
Pre-assignment Details: A total of 27 participants were enrolled in Parts 1 and 2 and 11 participants in Part 3. Part 2 was analyzed as a single arm as data was not collected for each dose level separately. The study was terminated as no participants in Part 3 showed a response and the potential risks outweighed potential benefit.
Groups:
- Part 1: Cohort 1 - 5 Micrograms/Kilogram/Dose (mcg/kg/Dose): Participants in this cohort received 5 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 for the first cycle of experimental drug followed by 9 days observation (Days 13 - 21) for a maximum of 6 cycles.
- Part 1: Cohort 2- 10 mcg/kg/Dose: Participants in this cohort received 10 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 for the first cycle of experimental drug followed by 9 days observation (Days 13 - 21) for a maximum of 6 cycles.
- Part 1: Cohort 3- 20 mcg/kg/Dose: Participants in this cohort received 20 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 for the first cycle of experimental drug followed by 9 days observation (Days 13 - 21) for a maximum of 6 cycles.
- Part 1: Cohort 4- 50 mcg/kg/Dose: Participants in this cohort received 50 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 for the first cycle of experimental drug followed by 9 days observation (Days 13 - 21) for a maximum of 6 cycles.
- Part 1: Cohort 5- 100 mcg/kg/Dose: Participants in this cohort received 100 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 for the first cycle of experimental drug followed by 9 days observation (Days 13 - 21) for a maximum of 6 cycles.
- Part 1: Cohort 6- 75 mcg/kg/Dose: Participants in this cohort received 75 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 of 21-Day cycle for up to 4 additional cycles to explore safety, tolerability and tumor response to repeat doses of MT-3724.
- Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose): Participants in this cohort either received 50 or 75 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 days of 21-Day cycle up to 4 additional cycles to explore safety, tolerability and tumor response to repeat doses of MT-3724.
- Part 3: MT-3724 was administered at a dose of 50μg/kg/dose via IV infusion for all participants
- Part 4: Participants in this arm were planned to receive all doses of MT-3724 as IV infusion over 1 hour in a 21-day cycle.
Period: Part 1 and 2 ( Up to Day 112)
Arm/Group | Part 1: Cohort 1 - 5 Micrograms/Kilogram/Dose (mcg/kg/Dose) | Part 1: Cohort 2- 10 mcg/kg/Dose | Part 1: Cohort 3- 20 mcg/kg/Dose | Part 1: Cohort 4- 50 mcg/kg/Dose | Part 1: Cohort 5- 100 mcg/kg/Dose | Part 1: Cohort 6- 75 mcg/kg/Dose | Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose) | Part 3 | Part 4
Started | 3 | 3 | 3 | 4 | 2 | 6 | 6 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 0 | 6 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: Part 3 (Up to Day 112)
Arm/Group | Part 1: Cohort 1 - 5 Micrograms/Kilogram/Dose (mcg/kg/Dose) | Part 1: Cohort 2- 10 mcg/kg/Dose | Part 1: Cohort 3- 20 mcg/kg/Dose | Part 1: Cohort 4- 50 mcg/kg/Dose | Part 1: Cohort 5- 100 mcg/kg/Dose | Part 1: Cohort 6- 75 mcg/kg/Dose | Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose) | Part 3 | Part 4
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Disease progression (radiographic per lugano) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0
Not completed — Clinical disease progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Period: Part 4 (Up to Day 112)
Arm/Group | Part 1: Cohort 1 - 5 Micrograms/Kilogram/Dose (mcg/kg/Dose) | Part 1: Cohort 2- 10 mcg/kg/Dose | Part 1: Cohort 3- 20 mcg/kg/Dose | Part 1: Cohort 4- 50 mcg/kg/Dose | Part 1: Cohort 5- 100 mcg/kg/Dose | Part 1: Cohort 6- 75 mcg/kg/Dose | Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose) | Part 3 | Part 4
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Part 2 was analyzed as a single arm as data was not collected for each dose level separately. As no participants from Part 3 had shown a response and as potential risks outweighed benefits, the study was terminated and no participants entered Part 4.
Groups:
- Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose): Participants in this cohort received 50 or 75 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 days of 21-Day cycle up to 4 additional cycles to explore safety, tolerability and tumor response to repeat doses of MT-3724.
- Part 3: All MT-3724 Treated Participants: MT-3724 was administered at a dose of 50µg/kg/dose via IV infusion for all participants
- Part 4: All MT-3724 Treated Participants: Participants in this arm were planned to receive all doses of MT-3724 as IV infusion over 1 hour in a 21-day cycle
- Total: Total of all reporting groups
Arm/Group | Part 1: Cohort 1 - 5 Micrograms/Kilogram/Dose (mcg/kg/Dose) | Part 1: Cohort 2- 10 mcg/kg/Dose | Part 1: Cohort 3- 20 mcg/kg/Dose | Part 1: Cohort 4- 50 mcg/kg/Dose | Part 1: Cohort 5- 100 mcg/kg/Dose | Part 1: Cohort 6- 75 mcg/kg/Dose | Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose) | Part 3: All MT-3724 Treated Participants | Part 4: All MT-3724 Treated Participants | Total
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 2 | 6 | 6 | 11 | 0 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.3 (6.43) | 70.7 (8.74) | 64.3 (14.01) | 57.8 (16.66) | 65.0 (4.24) | 67.2 (4.40) | 59.3 (10.58) | 57.5 (14.77) |  | 64.4 (5.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 3 | 1 | 4 | 5 | 3 |  | 20
  Male | 3 | 1 | 1 | 1 | 1 | 2 | 1 | 8 |  | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 3 | 3 | 2 | 2 | 5 | 6 | 11 |  | 34
  Asian | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 |  | 2
  Other | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities of a Single Cycle of MT-3724
Description: The MTD is defined to be the dose cohort below which participants experience dose-limiting toxicities during cycle 1. Dose-limiting toxicities were graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0
Time Frame: Days 1, 3, 5, 8, 10 and 12
Population: Safety Set comprises of all participants who received any amount of MT-3724
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 - 5 Micrograms/Kilogram/Dose (mcg/kg/Dose) | Part 1: Cohort 2- 10 mcg/kg/Dose | Part 1: Cohort 3- 20 mcg/kg/Dose | Part 1: Cohort 4- 50 mcg/kg/Dose | Part 1: Cohort 5- 100 mcg/kg/Dose | Part 1: Cohort 6- 75 mcg/kg/Dose
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 2 | 6
Participants | 0 | 0 | 0 | 0 | 2 | 0

2. Primary Outcome: Part 1 and 2: Maximum Observed Concentrations (Cmax) of MT-3274
Description: Blood samples were collected at indicated timepoints for the determination of Cmax of MT-3274.
Time Frame: Part 1 and 2 : Days 1, 3 and 12
Population: Pharmacokinetic Analysis Set (PAS). All subjects from the Safety Set with sufficient serum concentration data to determine the primary PK parameters. Only those participants with data available at specified timepoints were analyzed. Part 2 was analyzed as a single arm as data was not collected for each dose level separately.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Groups:
- Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose): Participants in this cohort received either 50 or 75 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 days of 21-Day cycle up to 4 additional cycles to explore safety, tolerability and tumor response to repeat doses of MT-3724.
Arm/Group | Part 1: Cohort 1 - 5 Micrograms/Kilogram/Dose (mcg/kg/Dose) | Part 1: Cohort 2- 10 mcg/kg/Dose | Part 1: Cohort 3- 20 mcg/kg/Dose | Part 1: Cohort 4- 50 mcg/kg/Dose | Part 1: Cohort 5- 100 mcg/kg/Dose | Part 1: Cohort 6- 75 mcg/kg/Dose | Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose)
Number analyzed (Participants) | 1 | 3 | 3 | 7 | 9 | 2 | 6
Nanograms per milliliter | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed)

3. Primary Outcome: Part 1 and 2: Time to Achieve Cmax (Tmax) of MT-3724
Description: Blood samples were collected at indicated timepoints for the determination of tmax.
Time Frame: Part 1 and 2: Days 1, 3 and 12
Population: Pharmacokinetic Analysis Set. Part 2 was analyzed as a single arm as data was not collected for each dose level separately.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Cohort 1 - 5 Micrograms/Kilogram/Dose (mcg/kg/Dose) | Part 1: Cohort 2- 10 mcg/kg/Dose | Part 1: Cohort 3- 20 mcg/kg/Dose | Part 1: Cohort 4- 50 mcg/kg/Dose | Part 1: Cohort 5- 100 mcg/kg/Dose | Part 1: Cohort 6- 75 mcg/kg/Dose | Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose)
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 2 | 6 | 6
Hours | NA [NA to NA] — Median and Full Range could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA [NA to NA] — Median and Full Range could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA [NA to NA] — Median and Full Range could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA [NA to NA] — Median and Full Range could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA [NA to NA] — Median and Full Range could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA [NA to NA] — Median and Full Range could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA [NA to NA] — Median and Full Range could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed)

4. Primary Outcome: Part 1 and 2: Area Under the Plasma Concentration Time Curve From 0 to 4 Hours (AUC [0-4]), AUC (0-infinity) and AUC From Dosing to Last Measurable Concentration (AUClast) of MT-3724
Description: Blood samples were collected at indicated timepoints for the determination of AUC (0-4), AUC (0-infinity) and AUClast.
Time Frame: Part 1 and 2: Days 1, 3 and 12
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/ml
Groups:
- Part 1: Cohort 2 - 10mcg/kg/Dose: Participants in this cohort received 10 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 for the first cycle of experimental drug followed by 9 days observation (Days 13 - 21) for a maximum of 6 cycles.
- Part 1: Cohort 3 - 20mcg/kg/Dose: Participants in this cohort received 20 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 for the first cycle of experimental drug followed by 9 days observation (Days 13 - 21) for a maximum of 6 cycles.
- Part 1: Cohort 4 - 50mcg/kg/Dose: Participants in this cohort received 50 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 for the first cycle of experimental drug followed by 9 days observation (Days 13 - 21) for a maximum of 6 cycles.
- Part 1: Cohort 5 - 100mcg/kg/Dose: Participants in this cohort received 100 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 for the first cycle of experimental drug followed by 9 days observation (Days 13 - 21) for a maximum of 6 cycles.
- Part 1: Cohort 6 - 75 mcg/kg/Dose: Participants in this cohort received 75 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 of 21-Day cycle for up to 4 additional cycles to explore safety, tolerability and tumor response to repeat doses of MT-3724.
Arm/Group | Part 1: Cohort 1 - 5 Micrograms/Kilogram/Dose (mcg/kg/Dose) | Part 1: Cohort 2 - 10mcg/kg/Dose | Part 1: Cohort 3 - 20mcg/kg/Dose | Part 1: Cohort 4 - 50mcg/kg/Dose | Part 1: Cohort 5 - 100mcg/kg/Dose | Part 1: Cohort 6 - 75 mcg/kg/Dose | Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose)
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 2 | 6 | 6
h*ng/ml
  AUC (0-4) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed)
  AUC (0-infinity) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed)
  AUClast | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed)

5. Primary Outcome: Part 1 and 2: Half Life (t1/2) of MT-3724
Description: Blood samples were collected at indicated timepoints for the analysis of t1/2 of MT-3724.
Time Frame: Part 1 and 2: Days 1, 3 and 12
Population: Pharmacokinetic Analysis Set. Part 2 was analyzed as a single-arm as data was not collected for each dose level separately.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Groups:
- Part 1: Cohort 1: 5 Micrograms/Kilograms/Dose/Day: Participants in this cohort received 5 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 of 21-Day cycle for up to 4 additional cycles to explore safety, tolerability and tumor response to repeat doses of MT-3724.
- Part 1: Cohort 2: 10 mcg/kg/Dose/Day: Participants in this cohort received 10 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 of 21-Day cycle for up to 4 additional cycles to explore safety, tolerability and tumor response to repeat doses of MT-3724.
- Part 1: Cohort 3: 20 mcg/kg/Dose/Day: Participants in this cohort received 20 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 of 21-Day cycle for up to 4 additional cycles to explore safety, tolerability and tumor response to repeat doses of MT-3724.
- Part 1: Cohort 4: 50 mcg/kg/Dose/Day: Participants in this cohort received 50 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 of 21-Day cycle for up to 4 additional cycles to explore safety, tolerability and tumor response to repeat doses of MT-3724.
- Part 1: Cohort 5: 100 mcg/kg/Dose/Day: Participants in this cohort received 100 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 of 21-Day cycle for up to 4 additional cycles to explore safety, tolerability and tumor response to repeat doses of MT-3724.
- Part 1: Cohort 6: 75 mcg/kg/Dose/Day: Participants in this cohort received 75 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 of 21-Day cycle for up to 4 additional cycles to explore safety, tolerability and tumor response to repeat doses of MT-3724.
Arm/Group | Part 1: Cohort 1: 5 Micrograms/Kilograms/Dose/Day | Part 1: Cohort 2: 10 mcg/kg/Dose/Day | Part 1: Cohort 3: 20 mcg/kg/Dose/Day | Part 1: Cohort 4: 50 mcg/kg/Dose/Day | Part 1: Cohort 5: 100 mcg/kg/Dose/Day | Part 1: Cohort 6: 75 mcg/kg/Dose/Day | Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose)
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 2 | 6 | 6
Hour | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed)

6. Primary Outcome: Part 1 and 2: Volume of Distribution (Vz) of MT-3724
Description: Blood samples were collected at indicated timepoints for the analysis of Vz of MT-3724.
Time Frame: Part 1 and 2: Days 1, 3 and 12
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Groups:
- Part 1: Cohort 1: 5 Micrograms/Kilograms/Dose/Day: Participants in this cohort received 5 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 for the first cycle of experimental drug followed by 9 days observation (Days 13 - 21) for a maximum of 6 cycles.
- Part 1: Cohort 2: 10 mcg/kg/Dose/Day: Participants in this cohort received 10 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 for the first cycle of experimental drug followed by 9 days observation (Days 13 - 21) for a maximum of 6 cycles.
- Part 1: Cohort 3: 20 mcg/kg/Dose/Day: Participants in this cohort received 20 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 for the first cycle of experimental drug followed by 9 days observation (Days 13 - 21) for a maximum of 6 cycles.
- Part 1: Cohort 4: 50 mcg/kg/Dose/Day: Participants in this cohort received 50 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 for the first cycle of experimental drug followed by 9 days observation (Days 13 - 21) for a maximum of 6 cycles.
- Part 1: Cohort 5: 100 mcg/kg/Dose/Day: Participants in this cohort received 100 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 for the first cycle of experimental drug followed by 9 days observation (Days 13 - 21) for a maximum of 6 cycles.
- Part 1: Cohort 6: 75 mcg/kg/Dose/Day: Participants in this cohort received 75 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 for the first cycle of experimental drug followed by 9 days observation (Days 13 - 21) for a maximum of 6 cycles.
Arm/Group | Part 1: Cohort 1: 5 Micrograms/Kilograms/Dose/Day | Part 1: Cohort 2: 10 mcg/kg/Dose/Day | Part 1: Cohort 3: 20 mcg/kg/Dose/Day | Part 1: Cohort 4: 50 mcg/kg/Dose/Day | Part 1: Cohort 5: 100 mcg/kg/Dose/Day | Part 1: Cohort 6: 75 mcg/kg/Dose/Day | Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose)
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 2 | 6 | 6
Liters | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed)

7. Primary Outcome: Part 1 and 2: Clearance (CL) of MT-3724
Description: Blood samples were collected at indicated timepoints for the analysis of CL of MT-3724.
Time Frame: Part 1 and 2: Days 1, 3 and 12
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 1: Cohort 1: 5 Micrograms/Kilograms/Dose/Day | Part 1: Cohort 2: 10 mcg/kg/Dose/Day | Part 1: Cohort 3: 20 mcg/kg/Dose/Day | Part 1: Cohort 4: 50 mcg/kg/Dose/Day | Part 1: Cohort 5: 100 mcg/kg/Dose/Day | Part 1: Cohort 6: 75 mcg/kg/Dose/Day | Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose)
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 2 | 6 | 6
Liters per hour | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed)

8. Primary Outcome: Part 1 and 2: Absolute Values of Cluster of Differentiation 19 Plus (CD19+) for B-cell Lymphocytes
Description: CD19+ cells in the peripheral blood were counted as measures of malignant B-cells and were measured by flow cytometry. Flow cytometry is a technique for counting and examining microscopic particles with an electronic detection apparatus
Time Frame: Part 1 and 2: Cycle 1: Days 8 and 23; Cycle 3: Day1; Cycle 5: Day 1 and Day 120 (end of study)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^3 cells per microliter
Groups:
- Part 1: Cohort 6- 75 mcg/kg/Dose: Participants in this cohort received 75 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 for the first cycle of experimental drug followed by 9 days observation (Days 13 - 21) for a maximum of 6 cycles.
- Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose): Participants in this cohort received either 50 or 75 mcg/kg/dose/day on Days 1, 3, 5, 8, 10, and 12 for the first cycle of experimental drug followed by 9 days observation (Days 13 - 21) for a maximum of 6 cycles.
Arm/Group | Part 1: Cohort 1 - 5 Micrograms/Kilogram/Dose (mcg/kg/Dose) | Part 1: Cohort 2- 10 mcg/kg/Dose | Part 1: Cohort 3- 20 mcg/kg/Dose | Part 1: Cohort 4- 50 mcg/kg/Dose | Part 1: Cohort 5- 100 mcg/kg/Dose | Part 1: Cohort 6- 75 mcg/kg/Dose | Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose)
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 0 | 6 | 0
10^3 cells per microliter
  Cycle 1 Day 8: number analyzed (Participants) | 1 | 2 | 1 | 3 | 0 | 1 | 0
  Cycle 1 Day 8 | 114 (NA) — Mean and Standard Deviation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | 325 (NA) — Mean and Standard Deviation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | 244 (NA) — Mean and Standard Deviation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | 57.7 (91.166) |  | 126 (NA) — NA indicates standard deviation could not be calculated for a single participant |
  Cycle 1 Day 23: number analyzed (Participants) | 1 | 2 | 1 | 0 | 0 | 1 | 0
  Cycle 1 Day 23 | 143 (NA) — Mean and Standard Deviation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | 104 (NA) — Mean and Standard Deviation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | 131 (NA) — Mean and Standard Deviation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) |  |  | 67.0 (NA) — NA indicates standard deviation could not be calculated for a single participant |
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 2 | 1 | 3 | 0 | 1 | 0
  Cycle 3 Day 1 | 67.0 (NA) — Mean and Standard Deviation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | 134 (NA) — Mean and Standard Deviation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | 60.0 (NA) — Mean and Standard Deviation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | 1170 (1965.6) |  | 34.0 (NA) — NA indicates standard deviation could not be calculated for a single participant |
  Cycle 5 Day 1: number analyzed (Participants) | 1 | 2 | 1 | 2 | 0 | 1 | 0
  Cycle 5 Day 1 | 132 (NA) — Mean and Standard Deviation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | 180 (NA) — Mean and Standard Deviation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | 53.0 (NA) — Mean and Standard Deviation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | 26.0 (31.1127) |  | 39.0 (NA) — NA indicates standard deviation could not be calculated for a single participant |
  Day 120 (End of study): number analyzed (Participants) | 1 | 2 | 1 | 3 | 0 | 1 | 0
  Day 120 (End of study) | 79.0 (NA) — Mean and Standard Deviation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | 184 (NA) — Mean and Standard Deviation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | 49.0 (NA) — Mean and Standard Deviation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | 22.87 (18.17) |  | 44.0 (NA) — NA indicates standard deviation could not be calculated for a single participant |

9. Primary Outcome: Part 1 and 2: Number of Participants With Positive Anti-drug Antibody (ADA) Confirmed
Description: Blood samples were collected to analyze the presence of ADA that bind MT-3724. Number of participants with positive ADA confirmed has been presented.
Time Frame: Part 1 and 2: Cycle 1, Day 23; Cycle 2, Day 1; Cycle 3, Day 1; Cycle 4, Day 1; Cycle 5, Day 1 and Day 120 (end of study)
Population: Pharmacokinetic Analysis Set. Only those participants with data available at specified time points has been presented. Part 2 was analyzed as a single arm as data was not collected for each dose level separately.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 - 5 Micrograms/Kilogram/Dose (mcg/kg/Dose) | Part 1: Cohort 2- 10 mcg/kg/Dose | Part 1: Cohort 3- 20 mcg/kg/Dose | Part 1: Cohort 4- 50 mcg/kg/Dose | Part 1: Cohort 5- 100 mcg/kg/Dose | Part 1: Cohort 6- 75 mcg/kg/Dose | Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose)
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 2 | 6 | 0
Participants
  Cycle 1 Day 23: number analyzed (Participants) | 1 | 3 | 2 | 3 | 1 | 5 | 0
  Cycle 1 Day 23 | 0 | 3 | 1 | 1 | 0 | 1 |
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 3 | 2 | 4 | 0 | 6 | 0
  Cycle 2 Day 1 | 0 | 3 | 1 | 4 | 0 | 2 |
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 2 | 1 | 3 | 0 | 1 | 0
  Cycle 3 Day 1 | 0 | 2 | 1 | 2 | 0 | 1 |
  Cycle 4 Day 1: number analyzed (Participants) | 1 | 2 | 1 | 3 | 0 | 1 | 0
  Cycle 4 Day 1 | 1 | 2 | 1 | 2 | 0 | 1 |
  Cycle 5 Day 1: number analyzed (Participants) | 1 | 2 | 1 | 2 | 0 | 1 | 0
  Cycle 5 Day 1 | 1 | 2 | 1 | 1 | 0 | 1 |
  Day 120 (end of study): number analyzed (Participants) | 3 | 2 | 2 | 4 | 1 | 5 | 0
  Day 120 (end of study) | 2 | 2 | 1 | 4 | 0 | 3 |

10. Primary Outcome: Part 3: Number of Participants Reporting Serious Treatment-emergent Adverse Events (TEAEs) and Non-serious TEAEs
Description: An adverse event is any untoward medical occurrence or clinical investigation in a participant administered a pharmaceutical product(s) and which does not necessarily have to have a causal relationship with this experimental treatment(s). SAE is any untoward medical occurrence, at any dose; is fatal or life-threatening, is life-threatening, results in permanently disabling; results in unplanned in-patient hospitalization or prolongation of existing hospitalization; results in a congenital abnormality or birth defect; important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when based upon appropriate medical judgment, they may jeopardize the participant or may require medical or surgical intervention.
Time Frame: Up to Day 45
Population: Safety Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 11
Participants
  Serious TEAEs | 3
  Non-serious TEAEs | 11

11. Primary Outcome: Part 3: Number of Participants With Clinically Significant Laboratory Parameters
Description: Blood samples were collected at indicated timepoints for the analysis of laboratory parameters.
Time Frame: Up to Day 45
Population: Safety Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 11
Participants | 0

12. Primary Outcome: Part 3: Number of Participants With Clinically Significant Electrocardiogram (ECG) Values
Description: Standard resting 12-lead ECG assessments was performed after the participant has rested quietly for at least 5 minutes in supine or semi-recumbent position.
Time Frame: Up to Day 26
Population: Safety Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 11
Participants | 0

13. Primary Outcome: Part 3: Number Participants With Clinically Significant Vital Signs
Description: Vital signs including systolic and diastolic blood pressure, respiratory rate, heart rate and body temperature were assessed at indicated time points.
Time Frame: Up to Day 45
Population: Safety Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 11
Participants | 0

14. Primary Outcome: Part 3: Number of Participants With Clinically Significant Physical Findings
Description: Physical examination was performed by a physician or a qualified delegate at the investigating site.
Time Frame: Up to Day 26
Population: Safety Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 11
Participants | 2

15. Primary Outcome: Part 4: Overall Response Rate (ORR) in MT-3724 Treated Participants With Relapsed or Refractory DLBCL
Description: Overall response rate is defined as the percentage of participants with either a CR or a PR as determined by independent, blinded central review.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

16. Secondary Outcome: Part 1 and 2: Number of Participants Reporting Worst Case Serious Treatment Emergent Adverse Events (TEAEs) and Non-serious TEAEs
Description: as for outcome 10
Time Frame: Up to Day 45
Population: Safety Set comprises of all participants who received any amount of MT-3724. Part 2 was analyzed as a single arm as data was not collected for each dose level separately.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 - 5 Micrograms/Kilogram/Dose (mcg/kg/Dose) | Part 1: Cohort 2- 10 mcg/kg/Dose | Part 1: Cohort 3- 20 mcg/kg/Dose | Part 1: Cohort 4- 50 mcg/kg/Dose | Part 1: Cohort 5- 100 mcg/kg/Dose | Part 1: Cohort 6- 75 mcg/kg/Dose | Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose)
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 2 | 6 | 6
Participants
  Serious TEAEs | 1 | 0 | 2 | 4 | 2 | 3 | 2
  Non-serious TEAEs | 3 | 3 | 3 | 4 | 2 | 6 | 6

17. Secondary Outcome: Part 3: ORR in MT-3724 Treated Participants With Relapsed or Refractory DLBCL by the Lugano Classification for Lymphoma
Description: Overall response rate is defined as the percentage of participants with either a complete response (CR) or a partial response (PR) as determined by independent, blinded central review board.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination.
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

18. Secondary Outcome: Part 3: ORR in MT-3724 Treated Participants With Relapsed or Refractory DLBCL
Description: Overall response rate is defined as the percentage of participants with either a CR or a PR as determined by investigator assessment.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

19. Secondary Outcome: Part 3: Duration of Tumor Response (DOR) in MT-3724 Treated Participants With Relapsed or Refractory DLBCL
Description: DOR defined as time from initial documentation of tumor response (CR or PR) to disease progression.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

20. Secondary Outcome: Part 3: Disease Control Rate (DCR) in MT-3724 Treated Participants With Relapsed or Refractory DLBCL
Description: DCR defined as percentage of participants who have achieved CR, PR and stable disease.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

21. Secondary Outcome: Part 3: Cmax of MT-3724 Monotherapy in Participants With Relapsed or Refractory DLBCL
Description: Blood samples were planned to be collected at indicated timepoints for the analysis of Cmax of MT-3724 monotherapy.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

22. Secondary Outcome: Part 3: Tmax of MT-3724 Monotherapy in Participants With Relapsed or Refractory DLBCL
Description: Blood samples were planned to be collected at indicated timepoints for the analysis of tmax of MT-3724 monotherapy.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

23. Secondary Outcome: Part 3: AUC (0-4), AUC (0-infinity) and AUClast of MT-3724 Monotherapy in Participants With Relapsed or Refractory DLBCL
Description: Blood samples were planned to be collected at indicated timepoints for the analysis of AUC (0-4), AUC (0-infinity) and AUClast of MT-3724 monotherapy.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

24. Secondary Outcome: Part 3: t1/2 of MT-3724 Monotherapy in Participants With Relapsed or Refractory DLBCL
Description: Blood samples were planned to be collected at indicated timepoints for the analysis of t1/2 of MT-3724 monotherapy.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

25. Secondary Outcome: Part 3: Vz of MT-3724 Monotherapy in Participants With Relapsed or Refractory DLBCL
Description: Blood samples were planned to be collected at indicated timepoints for the analysis of Vz of MT-3724 monotherapy.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

26. Secondary Outcome: Part 3: CL of MT-3724 Monotherapy in Participants With Relapsed or Refractory DLBCL
Description: Blood samples were planned to be collected at indicated timepoints for the analysis of CL of MT-3724 monotherapy
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

27. Secondary Outcome: Part 3: PD of MT-3724 Measured by B-cell Count in Participants With Relapsed or Refractory DCBCL
Description: Pharmacodynamics of MT-3724 was planned to be measured by B-cell count in participants with relapsed of refractory DCBCL using flow cytometry.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

28. Secondary Outcome: Part 3: PD of MT-3724 Measured by Immunophenotyping in Participants With Relapsed or Refractory DCBCL
Description: Pharmacodynamics of MT-3724 was planned to be measured by immunophenotyping in participants with relapsed of refractory DCBCL using flow cytometry.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

29. Secondary Outcome: Part 3: PD of MT-3724 Measured by Circulating Immunoglobulins in Participants With Relapsed or Refractory DCBCL
Description: Pharmacodynamics of MT-3724 was planned to be measured by circulating immunoglobulins in participants with relapsed of refractory DCBCL.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

30. Secondary Outcome: Part 3: Number of Participants With ADA When Treated With MT-3724
Description: Blood samples were planned to be collected to analyze the presence of ADA that bind MT-3724.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 3: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

31. Secondary Outcome: Part 4: DOR in MT-3724 Treated Participants With Relapsed or Refractory DLBCL
Description: Duration of response was defined as the time from the first occurrence of either complete or partial response to first documented evidence of disease recurrence or progression. Participants without evidence of progression were planned to be censored at time of last disease assessment. Only responders (CR or PR) were planned to be included for this analysis.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

32. Secondary Outcome: Part 4: Number of Participants Reporting Serious Treatment-emergent Adverse Events (TEAEs) and Non-serious TEAEs
Description: as for outcome 10
Time Frame: Up to Day 45
Population: Safety Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

33. Secondary Outcome: Part 4: Number of Participants With SAEs
Description: A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, any other situation such as important medical events according to medical or scientific judgement or is associated with liver injury and impaired liver function.
Time Frame: Up to Day 45
Population: Safety Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

34. Secondary Outcome: Part 4: Number of Participants With Clinically Significant Laboratory Parameters
Description: Blood samples were planned to be collected for the analysis of laboratory parameters.
Time Frame: Up to Day 45
Population: Safety Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

35. Secondary Outcome: Part 4: Number Participants With Clinically Significant Vital Signs
Description: Vital signs parameters including systolic and diastolic blood pressure, heart rate, respiration rate, body temperature and body weight were planned to be analyzed.
Time Frame: Up to Day 45
Population: Safety Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

36. Secondary Outcome: Part 4: Number of Participants With Clinically Significant ECG Values
Description: Standard resting 12-lead ECG assessments was planned to be performed after the participant has rested quietly for at least 5 minutes in supine or semi-recumbent position.
Time Frame: Up to Day 26
Population: Safety Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

37. Secondary Outcome: Part 4: Number of Participants With Adverse Events Suggestive of Cardiotoxicity
Description: Number of participants with any adverse events leading to cardiotoxicity when treated with MT-3724 was planned to be analyzed.
Time Frame: Up to Day 26
Population: Safety Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

38. Secondary Outcome: Part 4: ORR in MT-3724 Treated Participants With Relapsed or Refractory DLBCL
Description: Overall response rate was defined as the percentage of participants with either a CR or a PR as determined by investigator assessment.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

39. Secondary Outcome: Part 4: DCR in MT-3724 Treated Participants With Relapsed or Refractory DLBCL
Description: DCR was defined as percentage of participants who has achieved CR, PR and stable disease.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

40. Secondary Outcome: Part 4: Progression-free Survival (PFS) in MT-3724 Treated Participants With Relapsed or Refractory DLBCL
Description: Progression-free survival was defined as the time from study enrollment to the earliest date of disease progression or death from any cause.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

41. Secondary Outcome: Part 4: Overall Survival (OS) in MT-3724 Treated Participants With Relapsed or Refractory DLBCL
Description: Overall survival was defined as the time from study enrollment to death from any cause.
Time Frame: Up to Day 45
Population: Full Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

42. Secondary Outcome: Part 4: Cmax of MT-3724 Monotherapy in Participants With Relapsed or Refractory DLBCL
Description: Blood samples were planned to be collected at indicated timepoints for the analysis of Cmax of MT-3724 monotherapy.
Time Frame: Up to Day 45
Population: Pharmacokinetic Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

43. Secondary Outcome: Part 4: Tmax of MT-3724 Monotherapy in Participants With Relapsed or Refractory DLBCL
Description: Blood samples were planned to be collected at indicated timepoints for the analysis of Tmax of MT-3724 monotherapy.
Time Frame: Up to Day 45
Population: Pharmacokinetic Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

44. Secondary Outcome: Part 4: AUC (0-4), AUC (0-infinity) and AUClast of MT-3724 Monotherapy in Participants With Relapsed or Refractory DLBCL
Description: as for outcome 23
Time Frame: Up to Day 45
Population: Pharmacokinetic Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

45. Secondary Outcome: Part 4: t1/2 of MT-3724 Monotherapy in Participants With Relapsed or Refractory DLBCL
Description: Blood samples were planned to be collected at indicated timepoints for the analysis of t1/2 of MT-3724 monotherapy.
Time Frame: Up to Day 45
Population: Pharmacokinetic Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

46. Secondary Outcome: Part 4: Vz of MT-3724 Monotherapy in Participants With Relapsed or Refractory DLBCL
Description: Blood samples were planned to be collected at indicated timepoints for the analysis of Vz of MT-3724 monotherapy.
Time Frame: Up to Day 45
Population: Pharmacokinetic Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

47. Secondary Outcome: Part 4: CL of MT-3724 Monotherapy in Participants With Relapsed or Refractory DLBCL
Description: Blood samples were planned to be collected at indicated timepoints for the analysis of CL of MT-3724 monotherapy.
Time Frame: Up to Day 45
Population: Pharmacokinetic Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

48. Secondary Outcome: Part 4: PD of MT-3724 Measured by B-cell Count in Participants With Relapsed or Refractory DCBCL
Description: as for outcome 27
Time Frame: Up to Day 45
Population: Pharmacokinetic Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

49. Secondary Outcome: Part 4: PD of MT-3724 Measured by Immunophenotyping in Participants With Relapsed or Refractory DCBCL
Description: as for outcome 28
Time Frame: Up to Day 45
Population: Pharmacokinetic Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

50. Secondary Outcome: Part 4: PD of MT-3724 Measured by Circulating Immunoglobulins in Participants With Relapsed or Refractory DCBCL
Description: as for outcome 29
Time Frame: Up to Day 45
Population: Pharmacokinetic Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

51. Secondary Outcome: Part 4: Number of Participants With ADA When Treated With MT-3724
Description: Blood samples were planned to be collected to analyze the presence of ADA that bind MT-3724.
Time Frame: Up to Day 45
Population: Pharmacokinetic Analysis Set. The data was not collected due to early study termination
Arm/Group | Part 4: All MT-3724 Treated Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Non-serious TEAEs and SAEs were collected up to Day 45.
Description: Non-serious TEAEs and SAEs were collected in Safety Set and categorized using Common Terminology Criteria for Adverse Events (CTCAE) grade (1 to 5) where each grade is classified as grade 1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threatening and grade 5=fatal. Number of participants with worst case grade >=3 TEAEs and non-serious TEAEs has been presented. Part 2 was analyzed as a single arm as data was not collected for each dose level separately.
Groups:
- Part 3: All MT-3724 Treated Participants: Participants in this arm received all doses of MT-3724 as IV infusion over 1 hour in a 21-day cycle
Arm/Group | Part 1: Cohort 1: 5 Micrograms/Kilograms/Dose/Day | Part 1: Cohort 2: 10 mcg/kg/Dose/Day | Part 1: Cohort 3: 20 mcg/kg/Dose/Day | Part 1: Cohort 4: 50 mcg/kg/Dose/Day | Part 1: Cohort 5: 100 mcg/kg/Dose/Day | Part 1: Cohort 6: 75 mcg/kg/Dose/Day | Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose) | Part 3: All MT-3724 Treated Participants | Part 4: All MT-3724 Treated Participants
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 1/4 | 0/2 | 0/6 | 0/6 | 1/11 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 2/3 | 4/4 | 2/2 | 3/6 | 2/6 | 3/11 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 4/4 | 2/2 | 6/6 | 6/6 | 11/11 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Cohort 1: 5 Micrograms/Kilograms/Dose/Day (N=3) | Part 1: Cohort 2: 10 mcg/kg/Dose/Day (N=3) | Part 1: Cohort 3: 20 mcg/kg/Dose/Day (N=3) | Part 1: Cohort 4: 50 mcg/kg/Dose/Day (N=4) | Part 1: Cohort 5: 100 mcg/kg/Dose/Day (N=2) | Part 1: Cohort 6: 75 mcg/kg/Dose/Day (N=6) | Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose) (N=6) | Part 3: All MT-3724 Treated Participants (N=11) | Part 4: All MT-3724 Treated Participants (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Superinfection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Cohort 1: 5 Micrograms/Kilograms/Dose/Day (N=3) | Part 1: Cohort 2: 10 mcg/kg/Dose/Day (N=3) | Part 1: Cohort 3: 20 mcg/kg/Dose/Day (N=3) | Part 1: Cohort 4: 50 mcg/kg/Dose/Day (N=4) | Part 1: Cohort 5: 100 mcg/kg/Dose/Day (N=2) | Part 1: Cohort 6: 75 mcg/kg/Dose/Day (N=6) | Part 2: Cohort 7- MTD Expansion Cohort (50 or 75 mcg/kg/Dose) (N=6) | Part 3: All MT-3724 Treated Participants (N=11) | Part 4: All MT-3724 Treated Participants (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Retinal exudates (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Asthenia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 1 | 3 | 3 | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Reflux gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Anemia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 2 | 1 | 0 | 2 | 2 | 2 | 0
Infusion site irritation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Local swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Muscular weakness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Oedema peripheral (General disorders) | 1 | 3 | 0 | 4 | 1 | 4 | 3 | 4 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 1 | 3 | 1 | 6 | 0
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyoderma (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood chloride increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood lactic acid increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 4 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 2 | 2 | 3 | 7 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0
Horner's syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphoria (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 3 | 2 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT02361346/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT02361346/SAP_001.pdf